CLINICAL TRIAL: NCT02507310
Title: Influence of Ambient Temperature on Office Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Molly C. Bernhard, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: X141114013
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Environment

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Control (Active Comparator): The room will be kept at 18-20 degrees Celsius. This is within the human thermoneutral zone. It will serve as the control condition.
  Interventions: Other: thermostat
- Warm Environment (Experimental): The room will be kept at 25-27 degrees Celsius. This is above the human thermoneutral zone. This will serve as the experimental condition.
  Interventions: Other: thermostat

INTERVENTIONS:
Other: thermostat — ambient temperature as modified by thermostat
  Other Names: Environmental

SUMMARY:
Based on preliminary data and previous studies, we hypothesize that the ambient temperature experienced by an individual influences his or her food intake. Specifically, exposure to temperatures above the thermoneutral zone (TNZ) will decrease consumption in young adults in a sedentary situation. Researchers will execute a crossover randomized control trial specifically testing thermal exposure and its effect on individual female's food consumption.

DETAILED DESCRIPTION:
Participants will receive and wear a t-shirt. They will have a thermal image taken of the inner canthus of their eye and middle finger nail bed, representing a baseline of core and peripheral temperatures, respectively. They will also have their metabolic rate measured via a canopy hood method. At their initial visit, they will be randomized to either a colder environment (66-68°F) or a warmer environment (77-79°F) under the artifice of monitoring routine office work with abnormal temperature conditions. Their knowledge of the experiment will be limited until the end. They will experience this temperature while filling out paperwork and performing basic office tasks for a 7 hour work day. At the beginning and end of each day they will fill out a questionnaire on their appetite and thermal comfort. After the first 3.5 hours, another thermal image will be taken and the participant will be presented with lasagna and water and directed to eat at their leisure and subsequently finish the office tasks over the next 3.5 hours. A thermal image will be taken and metabolic rate will be assessed at the end of the day. Snacks will be available throughout the day. The participants will return approximately 1 week later to experience the other thermal environment following the same protocols. The participants will then be debriefed on the parameters of the experiment and body measurements will be taken at the end so as to prevent bias of the subject by limiting their food intake. We will quantify energy intake by weighing remaining food and comparing to known caloric content by weight from bomb calorimetry tests. The infrared thermal images will determine whether the temperatures experienced were extreme enough to initiate a change in thermoregulation.

ELIGIBILITY:
Inclusion Criteria:

Are you willing to have your height and weight taken? Are you willing and able to give informed consent? Are you able to communicate with the pertinent staff? Are you comfortable reading independently and answering a couple written questions related to the passage that you've read? Are you willing to sit in a small office with a closed door for an entire workday? Do you feel uncomfortable in confined spaces for extended periods of time?

Exclusion Criteria:

- Do you have any food allergy, including, but not limited to lactose or gluten intolerance? Do you have any religious affiliations that include specific food guidelines? Do you have any personal dietary restrictions, including but not limited to veganism? Have you participated in any weight-reduction program, weight-loss diet, or other special diet within the previous 3 months? Have you had weight loss or gain of >5% of body weight in the past 6 months for any reason except post-partum weight loss? Are you currently taking medication that suppresses or stimulates appetite or that affects body weight, including oral anti-diabetics medications? Do you have a history of prior surgical procedure for weight control or liposuction? Are you currently taking statins? Do you have high blood pressure (above 140 systolic, 90 diastolic)? Are you a current smoker or have you quit smoking less than 6 months prior?

Do you have any major disease, including:

* Active cancer or cancer requiring treatment in the past 2 years (except nonmelanoma skin cancer).
* Active or chronic infections, including self-reported HIV positivity and active tuberculosis.
* Active cardiovascular disease or event including hospitalization or therapeutic procedures for treatment of heart disease (e.g., coronary artery bypass, percutaneous transluminal coronary angioplasty) in the past 6 months; New York Heart Association Functional Class >2 with respect to congestive heart failure; stroke or transient ischemic attack in the past 6 months.
* Gastrointestinal disease, including self-reported chronic hepatitis or cirrhosis, any episode of alcoholic hepatitis or alcoholic pancreatitis within past year, inflammatory bowel disease requiring treatment in the past year, recent or significant abdominal surgery (e.g., gastrectomy).
* Active renal disease.
* Lung disease: chronic obstructive airway disease requiring use of oxygen.
* Diagnosed diabetes (type 1 or 2).
* Uncompensated or uncontrolled psychiatric disease (such as schizophrenia and bipolar disorder) that, in opinion of the investigators, would impede conduct of the trial or completion of procedures.

Do you have a history of or currently have an eating disorder? Have you ever been diagnosed with Raynaud's syndrome? Do you have another household member is a participant or staff member in the trial? Are you currently or do you anticipate participating in another intervention research project that would interfere with the intervention offered in the session? Are you willing to accept condition that you are randomized to? Are you currently taking antidepressant, steroid, or thyroid medication, unless dosage has been stable for at least 6 months? Do you have a recent or ongoing problem with drug abuse or addiction? Do you on average consume 3 or more alcohol containing beverages daily? Have you consumed 7 or more alcoholic beverages within a 24-hr period in the past 12 months? Are you a student in the Environmental Health Science Department, Nutrition Sciences School, any student, trainee, or post-doctoral fellow who is directly or indirectly receiving funding from the Nutrition Obesity Research Center? Are you currently pregnant or less than 3 months post-partum? Are you currently nursing or within 6 weeks of having completed nursing? Do you anticipate a pregnancy between time of screening and session date? Are you willing to report possible or confirmed pregnancies promptly at the time of the session?

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
food intake (kg) | Two workdays

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham School of Public Health, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Richardson MB, Li P, Gohlke JM, Allison DB. Effects of Indoor Thermal Environment on Human Food Intake, Productivity, and Comfort: Pilot, Randomized, Crossover Trial. Obesity (Silver Spring). 2018 Dec;26(12):1826-1833. doi: 10.1002/oby.22328. Epub 2018 Nov 14. PMID 30426700